CLINICAL TRIAL: NCT06023927
Title: Obstructive Sleep Apnea as a Risk Factor for Normal Tension Glaucoma and a Crucial Step in Preventing Blindness
Status: Not yet recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0958-MEETH
Record Dates: First submitted 2023-04-12; First posted 2023-09-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Normal Tension Glaucoma; Obstructive Sleep Apnea
Keywords: Glaucoma, obstructive sleep apnea Syndrome
MeSH Terms: conditions — Low Tension Glaucoma; Sleep Apnea, Obstructive; Glaucoma | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Newly-diagnosed mild OSA - initiating CPAP treatment: Subjects with newly-diagnosed mild obstructive sleep apnea being treated with CPAP undergoing clinical observation/diagnostic evaluation for detection and tracking of NTG.
  Interventions: Other: Clinical observation, diagnostic testing
- Newly-diagnosed moderate OSA - initiating CPAP treatment: Subjects with newly-diagnosed moderate obstructive sleep apnea being treated with CPAP undergoing clinical observation/diagnostic evaluation for detection and tracking of NTG.
  Interventions: Other: Clinical observation, diagnostic testing
- Newly-diagnosed severe OSA - initiating CPAP treatment: Subjects with newly-diagnosed severe obstructive sleep apnea being treated with CPAP undergoing clinical observation/diagnostic evaluation for detection and tracking of NTG.
  Interventions: Other: Clinical observation, diagnostic testing

INTERVENTIONS:
Other: Clinical observation, diagnostic testing — Glaucoma evaluation including structural and functional diagnostic testing at baseline and 3 subsequent follow-up visits over a period of 9 months

SUMMARY:
The purpose of this research study is to learn more about the relationship between Obstructive Sleep Apnea (OSA) and Normal Tension Glaucoma (NTG). OSA is a nighttime disorder of the upper airway that causes an intermittent lack of oxygen while sleeping. NTG is a type of glaucoma that occurs despite the normal intraocular pressure levels, making its detection more difficult. Left untreated, irreversible optic nerve damage and extensive vision loss can result. Previous research has shown some evidence between OSA and the development of NTG. The investigators are researching whether undergoing treatment for OSA would help to improve the vascular health to the retina, and in effect, improve the early signs of visual dysfunction seen with diagnostic testing.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of irreversible blindness worldwide. Normal tension glaucoma (NTG) is a challenging subtype in which progressive changes to the optic nerve and retinal ganglion cell (RGC) function occur despite normal intraocular pressures (IOP). In most types of glaucoma, elevated IOP is the major risk factor and a key target for medical therapy. The absence of IOP elevation in NTG poses diagnostic dilemmas and therapeutic challenges. The disease is often diagnosed late, with irreversible atrophic changes to the optic nerve and permanent loss of vision. These clinically manifested structural and functional changes seen on optical coherence tomography (OCT) and visual field (VF) tests are likely preceded by a subclinical stage at which RGCs become increasingly dysfunctional before dying.

Obstructive sleep apnea (OSA) is characterized by intermittent nocturnal upper airway collapse, leading to oxygen deprivation and hypoxemia. It is a common cause of daytime sleepiness and is associated with an increased likelihood of hypertension, cardiovascular disease, stroke, and diminished quality of life. Continuous Positive Airway Pressure (CPAP) therapy is an established treatment for moderate to severe OSA in which patients sleep with a special mask that helps to regulate inspiratory and expiratory flow, alleviating hypoxia.

The investigators hypothesize that eliminating the hypoxia induced by OSA could have a favorable effect on retinal blood flow, thereby reducing the likelihood of progressive RGC damage and dysfunction in subjects at risk for NTG. The investigators are proposing a prospective, longitudinal, non-randomized study to evaluate the role of innovative diagnostic technologies in the early detection of NTG, and to establish its association with OSA. Additionally, the investigators will monitor the effects of OSA treatment in preventing the development of the disease, or at least halting its progression. Special attention will be given to the sex differences in the analysis to recognize the substantial differences in OSA between men and women, as well as the prevalence of NTG in different OSA severity groups.

While under the care of a Sleep Medicine physician, newly diagnosed subjects with OSA interested in participating will be recruited from the Northwell sleep center. Prior to initiating continuous positive airway pressure therapy (CPAP), consented participants will be screened to satisfying the eligibility criteria, and undergo a complete ophthalmological exam. Functional and structural diagnostic testing will be performed to evaluate baseline measures, including visual field testing, OCT, pattern electroretinography (PERG) and optical coherence tomography-angiography (OCTA) testing. Using the American Association of sleep Medicine (AASM) criteria, 3 groups will be formed based on the apnea-hypopnea index (AHI). The severity of OSA is graded as mild (AHI<15), moderate (15<AHI<30), or severe (AHI>30). The Epworth questionnaire will be used as part of routine clinical care to monitor improvement or deterioration after treatment. Once the baseline ophthalmological exam has been performed, subjects will return to the sleep center to begin CPAP therapy for OSA. Three follow up ophthalmic exams will be performed at 3, 6, and 9 months after initiating CPA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed subjects with OSA that will undergo CPAP treatment.
* At least 21 years of age
* Best corrected vision of 20/40 or better, spherical Rx < ± 6.0 Diopter, and cylinder <-3.0D
* Ability to follow instructions, and intent to complete all study visits

Exclusion Criteria:

* High Rx >± 6.0D and cylinder > -3.0D
* Narrow angle glaucoma
* History of any of the following: severe eye trauma, ocular inflammation, previous intraocular surgery except for uncomplicated cataract extraction with posterior chamber intraocular lens implantation.
* Any medical or ocular condition which is not appropriate for participation in the trial (Diabetic retinopathy, and other retinal changes preventing reliable optic disc evaluation) Hypersensitivity to any component of altafluor benox

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Newly-diagnosed OSA patients that will undergo CPAP treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NTG | 2 years
  To determine the prevalence of normal tension glaucoma (NTG) in newly-diagnosed subjects with different stages of obstructive sleep apnea (mild, moderate, and severe)
Mean difference in diagnostic parameters at baseline | 2 years
  Mean difference in pattern electroretinogram (PERG) parameters (in millivolts) and optical coherence tomography angiography (OCTA) Vessel density (VD) measurements at baseline between the 3 OSA study groups (mild, moderate, and severe).Magnitude (mV), MagnitudeD (MagD) (mV), MagD/Mag ratio and VD (%) will be compared across 3 OSA groups
Mean change in diagnostic parameters at follow up intervals | 2 years
  Mean change in PERG parameters (in millivolt) and OCTA vessel density measurements (%) in each of the follow up visits compared to baseline
Two PERG devices will be compared in their ability to detect retinal ganglion cell dysfunction | 2 years
  Diopsys NOVA PERG parameters will be correlated with PERG SmartEP parameters (in millivolts)

SECONDARY OUTCOMES:
Incidence of NTG in female subjects | 2 years
  Incidence of NTG in female subjects
Correlation of polysomnography and Epworth Sleeping Scale measures with PERG (Mag,MagD in millivolts, MagD/Mag ratio)and OCTA VD (%) measurements | 2 years
  Correlation of day time sleepiness from the Epworth scale (in points), polysomnography measures (apnea-hypopnea Index, in events/hour, saturation of oxygen, SaO2 in %, ), with PERG Mag, MagD in mV, MagD/Mag ratio and OCTA VD (in %) measurements
Correlations between PERG parameters, Ocular Perfusion Pressure (OPP) and corneal hysteresis | 2 years
  Correlations between Mag, magD (in mV) and MagD/Mag ration, OPP measured by Falck device (mm Hg) , and corneal hysteresis (mm Hg), provided by ocular response analyzer, will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Manhattan Eye, Ear, & Throat Hospital, New York, New York, United States